CLINICAL TRIAL: NCT03405324
Title: Effect of the Transcranial Direct Current Stimulation (tDCS) of the Motor Cortex on Chemotherapy Induced Nausea and Vomiting in Breast Cancer Patients
Brief Title: Effect of tDCS of the Motor Cortex on Chemotherapy Induced Nausia and Vomiting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shereen Mamdouh (Other)
Responsible Party: Sponsor-Investigator, Shereen Mamdouh, Lecturer of anesthesia, ICU and pain relief, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 233
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: brain stimulation, tDCS, nausea and vomiting
MeSH Terms: conditions — Vomiting; Nausea | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active tDCS (Active Comparator): a single session over the primary motor cortex with constant current of 2mA intensity was applied for 20 minutes with a 5-second ramp phase at the beginning applied to the participant patient before chemotherapy .
  Interventions: Device: tDCS
- sham tDCS (Sham Comparator): a single session over the primary motor cortex with constant current of 2mA intensity was applied for 20 minutes with a 5-second ramp phase at the beginning applied to the participant patient before chemotherapy switched off after 30 second without the patient knowledge .
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: tDCS — a single session of tDCS over the primary motor cortex with constant current of 2mA intensity will be applied for 20 minutes with a 5-second ramp phase at the beginning.
  Arms: active tDCS
Device: sham tDCS — sham tDCS
  Arms: sham tDCS

SUMMARY:
this work is looking for the effect of tDCS of the motor cortex on the chemotherapy induced nausea and vomiting in cancer breast patients

DETAILED DESCRIPTION:
Chemotherapy has played an important role in improving patient outcomes in oncology and is a cornerstone of therapy for most patients with cancer. Of the adverse effects, none is more feared than chemotherapy-induced nausea and vomiting (CINV).

Nausea and vomiting can adversely affect patients' quality of life and make it difficult for them to perform their activities of daily living. Uncontrolled CINV can give rise to medical complications, including poor nutrition, dehydration, electrolyte imbalances, and physical and mental deterioration.The introduction and development of antiemetic drugs have significantly improved the ability of clinicians to control CINV. The mainstays of antiemetic therapy include serotonin (5-HT3) receptor antagonists (RAs) and neurokinin 1 (NK-1) RAs. Researchers and patients are seeking additional methods of controlling CINV, such as non-drug therapies. Transcranial direct current stimulation (tDCS) is a relatively simple technique requiring only a few parts.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer therapy receiving anthracyclin based adjuvant chemotherapy and prophylaxis against nausea and vomiting

Exclusion Criteria:

* patients with intracranial metallic devices or with pacemakers or any other device.
* patients with extensive myocardial ischemia
* patients known to have epilepsy patients refusal.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Cumulative of nausea scoring | the first 72 hours after the infusion of chemotherapy
  0=None
  1. Loss of appetite eout alternation in eating habits
  2. Dec. oral intake eout significant wgt loss, dehydration or malnutrion
  3. Iv fluids, tube feeding, TPN
  4. Life threatening consequence

SECONDARY OUTCOMES:
cumalative vomiting scoring | the first 72 hours after the infusion of chemotherapy
  0= None 1=1 episode in 24h 2= 2-5 episodes in 24h 3=More 6 episodes in 24h 4=Life threatening consequence

CONTACTS AND LOCATIONS:
Locations (1):
- South Egypt Cancer Institute, Asyut, Egypt

REFERENCES:
- [Derived] Kamal SM, Elhusseini NM, Sedik MF, Mohamad MF, Khedr EMH, Kotb HIM. Effect of Transcranial Direct Current Brain Stimulation of the Motor Cortex on Chemotherapy-Induced Nausea and Vomiting in Female Patients with Breast Cancer. Pain Med. 2022 Mar 2;23(3):571-578. doi: 10.1093/pm/pnab313. PMID 34677609